CLINICAL TRIAL: NCT01578863
Title: Predictors of Success in a Multidisciplinary Intervention Program for Obese Children and Adolescence
Brief Title: Predictors of Success in an Intervention Program for the Treatment of Childhood Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MeirMc009-12CTIL
Record Dates: First submitted 2012-03-15; First posted 2012-04-17 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2014-05

CONDITIONS: Childhood Obesity
Keywords: Childhood obesity; Adolescence; Predictors; Success; Intervention program
MeSH Terms: conditions — Pediatric Obesity | interventions — Exercise; Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intervention program (Active Comparator): 6 months intervention program to lose weight in obese children. Behavioral, emotional, physical, familial and demographic questioners will be fulfilled at the beginning and at the end of the program.
  Interventions: Other: Intervention program for obese children
- Untreated obese children (No Intervention): Behavioral, emotional, physical, familial and demographic questioners will be fulfilled twice in a 6 month program.
- Normal weight children (No Intervention): Behavioral, emotional, physical, familial and demographic questioners will fulfill twice in the 6 month period.

INTERVENTIONS:
Other: Intervention program for obese children — The program includes physical activity, nutrition intervention and behavioral treatment and lasts for 6 months. The aim of the program is to promote weight loss and physical activity and to promote future healthy lifestyle.
  Other Names: exercise, nutrition, behavioral
  Arms: Intervention program

SUMMARY:
The child health and sports center, at the Meir Medical Center, runs for over 10 years an intervention program to treat obese children. The program includes physical activity, nutritional intervention and behavioral treatment. A similar program exists in the nearby city of Hadera. The aim of the programs is to promote weight loss, encourage physical activity and modify behavior in order to get long term results. The aim of the present study is to try and identify the demographic and behavioral characteristics of children who succeed in the program.

ELIGIBILITY:
Inclusion Criteria:

* Obese / overweight children

Exclusion Criteria:

* Children that has an organic illness that cause obesity

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 176 (Actual)
Dates: Start 2012-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Characteristics of the children who succeed in the program | 6 Months
  We will use behavioral, emotional, physical, familial and demographic questionnaires to characterize the children taking part in the programs.
  The questionnaires: self-efficacy, motivation, depression, parenting style, demographic, environmental.Anthropometric and fitness measurements are performed on a monthly basis .

CONTACTS AND LOCATIONS:
Overall Officials: Dan Nemet, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel